CLINICAL TRIAL: NCT05112601
Title: A Randomized Phase II Trial of Nivolumab and Ipilimumab Compared to Nivolumab Monotherapy in Patients With Deficient Mismatch Repair System Recurrent Endometrial Carcinoma
Brief Title: Testing Nivolumab With or Without Ipilimumab in Deficient Mismatch Repair System (dMMR) Recurrent Endometrial Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-11881; NCI-2021-11881 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY025 (Other: NRG Oncology); NRG-GY025 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2021-11-06; First posted 2021-11-09 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-09

CONDITIONS: Endometrial Adenocarcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Dedifferentiated Carcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Mucinous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Endometrioid Adenocarcinoma; Recurrent Endometrial Carcinoma
MeSH Terms: conditions — Carcinoma, Endometrioid; Endometrial Neoplasms | interventions — Specimen Handling; Ipilimumab; CTLA-4 Antigen; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (nivolumab and ipilimumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1 of each cycle and ipilimumab IV over 90 minutes on day 1 of every other cycle. Cycles repeat every three weeks. Treatment with nivolumab and ipilimumab repeats for up to 8 cycles in the absence of disease progression, unacceptable toxicity, or CR. Patients then receive nivolumab alone on day 1 of each cycle. Cycles repeat every 4 weeks in the absence of disease progression, unacceptable toxicity, or CR.
  MAINTENANCE THERAPY: Patients achieving CR receive nivolumab for an additional 12 months in the absence of disease progression or unacceptable toxicity.
  Additionally, patients may optionally undergo collection of tissue samples on study as well as blood samples throughout the trial. Patients also undergo CT scan and/or MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Ipilimumab; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab
- Arm II (nivolumab) (Active Comparator): Patients receive nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for up to 8 cycles, then every 4 weeks thereafter in the absence of disease progression, unacceptable toxicity, or CR.
  MAINTENANCE THERAPY: Patients achieving CR receive nivolumab for an additional 12 months in the absence of disease progression or unacceptable toxicity.
  Additionally, patients may optionally undergo collection of tissue samples on study as well as blood samples throughout the trial. Patients also undergo CT scan and/or MRI throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Biological: Nivolumab

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of tissue and/or blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS 734016; BMS-734016; BMS734016; Ipilimumab Biosimilar CS1002; MDX 010; MDX-010; MDX-CTLA4; MDX010; Yervoy
  Arms: Arm I (nivolumab and ipilimumab)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo

SUMMARY:
This phase II trial tests whether the combination of nivolumab and ipilimumab is better than nivolumab alone to shrink tumors in patients with deficient mismatch repair system (dMMR) endometrial carcinoma that has come back after a period of time during which the cancer could not be detected (recurrent). Deoxyribonucleic acid (DNA) mismatch repair (MMR) is a system for recognizing and repairing damaged DNA. In 2-3% of endometrial cancers this may be due to a hereditary condition resulted from gene mutation called Lynch Syndrome (previously called hereditary nonpolyposis colorectal cancer or HNPCC). MMR deficient cells usually have many DNA mutations. Tumors that have evidence of mismatch repair deficiency tend to be more sensitive to immunotherapy. There is some evidence that nivolumab with ipilimumab can shrink or stabilize cancers with deficient mismatch repair system. However, it is not known whether this will happen in endometrial cancer; therefore, this study is designed to answer that question. Monoclonal antibodies, such as nivolumab and ipilimumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving nivolumab in combination with ipilimumab may be better than nivolumab alone in treating dMMR recurrent endometrial carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess efficacy in terms of progression-free survival (PFS) for immunotherapy with dual immune checkpoint blockade (nivolumab/ipilimumab) versus (vs.) monotherapy (nivolumab) in patients with recurrent mismatch repair (MMR) deficient endometrial carcinoma with measurable or non-measurable (detectable) disease.

SECONDARY OBJECTIVES:

I. To evaluate the overall survival (OS) as estimated from time of enrollment to last follow-up or death.

II. To evaluate the objective response rate by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in those with measurable disease at start of treatment.

III. To evaluate progression-free survival at 6 months. IV. To evaluate the nature, frequency and degree of toxicity as assessed by the Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

V. To evaluate PFS and objective response rate in patients with prior anti-PD1/PDL1 therapy and compare efficacy of dual immune checkpoint inhibition vs. anti-PD1 monotherapy.

OUTLINE: Patients are randomized into 1 of 2 arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes on day 1 of each cycle and ipilimumab IV over 90 minutes on day 1 of every other cycle. Cycles repeat every three weeks. Treatment with nivolumab and ipilimumab repeats for up to 8 cycles in the absence of disease progression, unacceptable toxicity, or complete response (CR). Patients then receive nivolumab alone on day 1 of each cycle. Cycles repeat every 4 weeks in the absence of disease progression, unacceptable toxicity, or CR.

ARM II: Patients receive nivolumab IV over 30 minutes on day 1 of each cycle. Treatment repeats every 3 weeks for up to 8 cycles, then every 4 weeks thereafter in the absence of disease progression, unacceptable toxicity, or CR.

MAINTENANCE THERAPY: Patients achieving CR on Arm I or II receive nivolumab for an additional 12 months in the absence of disease progression or unacceptable toxicity.

Additionally, all patients may optionally undergo collection of tissue samples on study as well as blood samples throughout the trial. All patients also undergo computed tomography (CT) scan and/or magnetic resonance imaging (MRI) throughout the trial.

Patients are followed every 3 months for 2 years, and then, every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with measurable or non-measurable (detectable) recurrent endometrial cancer
* Measurable disease will be defined and monitored by RECIST v 1.1. Measurable disease is defined per RECIST 1.1 criteria as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by computed tomography (CT) or magnetic resonance imaging (MRI). Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Non-measurable (detectable) disease in a patient is defined in this protocol per RECIST 1.1 criteria as one who does not have measurable disease but has at least one of the following conditions:

  * All other lesions (or sites of disease), including small lesions (longest diameter <10 mm or pathological lymph nodes with >= 10 to < 15 mm short axis), are considered non-measurable disease
  * Ascites and/or pleural effusion attributed to tumor
  * Solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions
* Patients must have endometrial cancer with deficient mismatch repair system. All patients must have institutional immunohistochemistry (IHC) and/or microsatellite instability (MSI) testing to determine mismatch repair (MMR) status. MMR deficiency is defined as lack of expression of one or more mismatch repair proteins (MLH1, PMS2, MSH2, MSH6, EPCAM) by immunohistochemistry and/or presence of microsatellite instability high using the National Cancer Institute (NCI)-5plex and Promega v1.2 assays, or institutional standards (e.g. next-generation sequencing [NGS] panel)

  * Method(s) of detection of MMR deficiency will be recorded for each patient. An institutional pathology report, and additional reports if available, documenting these results must be submitted. Patients with "equivocal" results on MMR testing by immunohistochemistry may be eligible if they have documented evidence of microsatellite instability by MSI testing or by next generation sequencing assays. MMR testing by IHC may be used to resolve equivocal/indeterminate MSI results
* Histologic confirmation of the original primary tumor is required (submission of pathology report(s) is required). Patients with the following histologic types are eligible: Endometrioid adenocarcinoma, mucinous adenocarcinoma, dedifferentiated/undifferentiated carcinoma, clear cell adenocarcinoma, mixed epithelial carcinoma, adenocarcinoma not otherwise specified (N.O.S.)
* Patients may have received 1-2 prior lines of systemic therapy:

  * Prior anti-PD1/PD-L1 therapy is allowed if given in combination with chemotherapy or radiation therapy in adjuvant or primary metastatic/recurrent settings. Patients must have had a complete response and have disease progression/relapse with treatment-free interval of 12 months or more from last dose of therapy with immune check inhibition
* Patients may have received prior radiation therapy for treatment of endometrial cancer. Prior radiation therapy may have included pelvic radiation therapy, extended field pelvic/para aortic radiation therapy, intravaginal brachytherapy, and/or palliative radiation therapy. All radiation therapy must be completed at least 4 weeks prior to registration
* Patients may have received prior hormonal therapy for treatment of endometrial cancer. All hormonal therapy must be discontinued at least three weeks prior to registration
* Any other prior therapy directed at the malignant tumor including chemotherapy, targeted agents, biologic agents, immunologic agents, and any investigational agents, must be discontinued at least 4 weeks prior to registration (6 weeks for nitrosoureas or mitomycin C)
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Platelets >= 100,000/mcl
* Absolute neutrophil count (ANC) >= 1,500/mcl
* Creatinine =< 1.5 x institutional/laboratory upper limit of normal (ULN)
* Total serum bilirubin level =< 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level =<3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN
* Adequate oxygen saturation via pulse oximeter (CTCAE v.5.0 hypoxia < grade 2 within 28 days prior to registration)
* Thyroid-stimulating hormone (TSH) within normal limits (TSH < ULN allowed in euthyroid patients on thyroid replacement therapy). TSH testing is only required if clinically indicated
* Patients must have recovered from effects of recent surgery, radiotherapy or chemotherapy. At least 4 weeks must have elapsed since major surgery
* As clinically indicated, patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better and have a corrected QT (QTc) interval < 450 msec
* The effects of nivolumab, and ipilimumab on the developing human fetus are unknown. For this reason and because nivolumab and ipilimumab are known to be teratogenic, women of child-bearing potential (WOCBP) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for 5 months after the last dose of investigational drug. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab. Women must not be breastfeeding. Women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile) do not require contraception

  * WOCBP is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression and the patient is stable off steroids for at least one month
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information
* Patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible
* Patients with rheumatoid arthritis and other arthropathies, Sjogren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible

Exclusion Criteria:

* Patients with a diagnosis of endometrial serous carcinoma or carcinosarcoma
* Patients who received prior anti-PD1/PD-L1 therapy and had grade 3-4 or recurring grade 2 immune-related toxicities that led to dose delay or discontinuation of immunotherapy due to those toxicities
* Patients who received anti-CTLA-4 therapy or other immunotherapeutic agents
* Patients on chronic steroid therapy except those on replacement therapy at a daily dose of 10mg or less prednisone or equivalent
* Patients on immunosuppressive therapy, with the exception of:

  * Intra-nasal, inhaled, topical or local steroid injections
  * Premedication for hypersensitivity reaction
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
* Patients with known immune impairment who may be unable to respond to anti-CTLA-4 antibody
* Patients with uncontrolled intercurrent illness including, but not limited to: ongoing or active infection (except for uncomplicated urinary tract infection), interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Women who are pregnant or unwilling to discontinue nursing
* Prior therapy with CTLA-4 inhibitors, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, and/or ipilimumab including severe hypersensitivity reactions to any monoclonal antibody

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-06-02 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years after randomization
  The statistical test used for decision making is the stratified, standardized log-rank test (Z) based on PFS. For the safety lead-in analysis, the primary endpoint is the observation of at least one dose-limiting toxicity (DLT) in the first 3 cycles of treatment. Patients are classified as having a DLT in 3 cycles or receiving adequate treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years after randomization
  Will be assessed when the PFS data are mature. The null hypothesis will be that the hazard of death in regimen 1 is equal to the hazard of death in regimen 2. That is, Ho: HR = 1.00. The alternative will be that Ha: HR < 1.00 (regimen 1 to 2). The number of deaths is unknown.
Objective tumor response (ORR) | Up to 5 years after randomization
  Defined as the frequency of patients who have either a partial or complete response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. The number of patients with responses will be tabulated by the treatment they were randomized to. Fisher's Exact Test will be used to test the hypothesis that the probabilities of response in each arm is the same. ORR will be evaluated only in patients who had measurable disease per RECIST 1.1 before starting treatment.
Progression-free survival (PFS) at 6 months | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed at 6 months after randomization
  A patient who survives at least 6 months progression-free will be considered to have had a successful outcome. Those who progress or die within 6 months are considered treatment failures, and those who survive progression-free for less than 6 months will be considered to have an unknown outcome or indeterminate. If the patient's status cannot be determined, she will be moved to the "failure" status for analysis. Like tumor response, the hypothesis of equivalent probabilities will be assessed with Fisher's Exact Test.
Incidence of adverse events | Up to 5 years after randomization
  Will be assessed by Common Terminology Criteria for Adverse Events (CTCAE). Will be tabulated by frequency and severity by treatment regimen. The treatment regimens will be compared by classifying the toxicities as severe or not and tested for equivalent probabilities by Fisher's Exact Test or whether the estimated probabilities of severe toxicities diverge by more than 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Haider S Mahdi, Principal Investigator — NRG Oncology
Locations (121):
- United States (121):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - University of Illinois, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Intermountain Health West End Clinic, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Essentia Health Cancer Center-South University Clinic, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - UPMC Hillman Cancer Center at Butler Health System, Butler, Pennsylvania
  - UPMC Hillman Cancer Center - Passavant - Cranberry, Cranberry Township, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - IRMC Cancer Center, Indiana, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - UPMC Hillman Cancer Center - Part of Frick Hospital, Mount Pleasant, Pennsylvania
  - Arnold Palmer Cancer Center Medical Oncology Norwin, N. Huntingdon, Pennsylvania
  - UPMC Cancer Center-Natrona Heights, Natrona Heights, Pennsylvania
  - UPMC Hillman Cancer Center - New Castle, New Castle, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Cancer Center-Washington, Washington, Pennsylvania
  - UPMC West Mifflin-Cancer Center Jefferson, West Mifflin, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm